CLINICAL TRIAL: NCT07264491
Title: Clinical Performance of Full Coverage Hybrid Ceramic Crowns in the Aesthetic Zone: A Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karim Ahmed Awadallah Osman (Other)
Responsible Party: Sponsor-Investigator, Karim Ahmed Awadallah Osman, Lecturer, Fixed Prosthodontics Department, Faculty of Dentistry, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2025-05-26
Record Dates: First submitted 2025-06-11; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Dental Restoration Failure of Marginal Integrity; Poor Aesthetic of Existing Restoration of Tooth
Keywords: clinical outcome- hybrid ceramics- resin cements; full coverage- marginal discrepancy

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vita Enamic Hybrid Ceramic full coverage Crowns (Active Comparator): Polymer-infiltrated-ceramic-network material (Vita Enamic)
  Interventions: Other: Shofu HC Hard full coverage corwns
- Shofu Hard HC full coverage crowns (Experimental): highly esthetic ceramic-based restorative (hybrid ceramics) for milling into dental restorations using a dental CAD/CAM system.
  Interventions: Other: Vita Enamic full coverage crowns

INTERVENTIONS:
Other: Shofu HC Hard full coverage corwns — HC HARD hybrid ceramic crowns
  Arms: Vita Enamic Hybrid Ceramic full coverage Crowns
Other: Vita Enamic full coverage crowns — hybrid cermaics
  Arms: Shofu Hard HC full coverage crowns

SUMMARY:
Participants will receive high-quality dental restorations, installed and monitored by qualified dental professionals regular periodic follow up recalls will be assigned early detect any consequences free of charge repairs or remakes for any failed dental restorations this research will help in the improvement of the tested materials

DETAILED DESCRIPTION:
Direct benefit of the research to the human volunteer:

* Participants will receive high-quality dental restorations (hybrid ceramic full coverage restorations) fabricated using standardized protocols and materials.
* All participants will have their restorations placed by qualified dental professionals in a controlled clinical environment, ensuring proper technique and follow-up care.
* Participants will benefit from regular follow-up examinations at 6, 12, and 18 months, which allows for early detection and management of any potential issues with their restorations.
* Any issues or failures identified during the follow-up period will be documented and repaired at no additional cost to the participant.
* Participants will contribute to advancing dental knowledge regarding optimal hybrid ceramic materials, which may lead to improved treatment protocols and long-term outcomes for future dental patients.
* The research provides an opportunity for comprehensive oral health monitoring beyond just the restoration itself, potentially identifying other dental issues that might require attention.

The scientific interest and the desired public benefit of the research:

Scientific Interest

1. This research will help understanding the material-specific outcomes in terms of marginal adaptation, color match, retention, surface texture, and restoration failure
2. The study will contribute to the understanding of the relationship between laboratory findings and clinical outcomes for dental materials, particularly regarding hybrid ceramics.
3. The findings may generate evidence on the clinical effectiveness and long-term behavior of two hybrid ceramic materials
4. The research will provide long-term clinical data on modern dental materials, which is valuable for developing future materials and techniques.
5. The study evaluates how the properties of Beautilink SA self-adhesive resin cement interact with these crown materials to affect clinical outcomes, offering new insights into optimal cementation protocols.

Desired Public Benefits

1. Providing evidence-based guidance for dental practitioners regarding different hybrid ceramic blocks.
2. Providing clinicians with evidence-based guidance for selecting the most suitable hybrid ceramic material for full coverage crowns in the esthetic zone.
3. Enhancing the longevity of restorations by identifying bonding protocols less prone to debonding, which is identified as one of the most common failure modes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients requiring full coverage crowns in aesthetic zone
2. Age ≥ 21 years
3. Vital or endodontically treated teeth
4. Willing and able to provide written informed consent
5. Ability to attend all follow-up appointments
6. Adequate oral hygiene as determined by the investigator

Exclusion Criteria:

1. Patients with active periodontal disease (probing depth > 4mm, bleeding on probing)
2. Patients with parafunctional habits (e.g., bruxism confirmed by clinical examination)
3. Poor oral hygiene (plaque index > 30%)
4. Systemic diseases affecting treatment outcomes (e.g., uncontrolled diabetes, immunosuppression)
5. Known allergies to study materials (ceramic materials, or resin cement components)
6. Inability to comply with study requirements
7. Current participation in other dental clinical trials

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
marginal adaptation | from enrollment to the end of treatment at 18 months
  measurement of vertical and horizontal discrepancies at the margins of dental restorations

SECONDARY OUTCOMES:
Color match | from enrollment to the end of treatment at 18 months
  measurement of any mismatch in the color or translucency using Modified USPHS criteria

CONTACTS AND LOCATIONS:
Overall Officials: Reham Elbasty, MSC, PhD, Study Director — Cairo University
Locations (1):
- Faculty Of Dentistry, Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giordano, R. (2016). Materials for chairside CAD/CAM-produced restorations. Journal of the American Dental Association, 147(12), 972-980. https://doi.org/10.1016/j.adaj.2016.07.002 (Overview of hybrid ceramics used in CAD/CAM and their esthetic/mechanical advantages.)